CLINICAL TRIAL: NCT01090180
Title: Extinction of Fear Memories With Glucocorticoids in Veterans With PTSD
Acronym: VA CORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D6902-R; 09-052 (Other: IRB protocol number)
Record Dates: First submitted 2010-03-15; First posted 2010-03-19 (Estimated); Results first posted 2016-11-25 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-10

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; combat; stress disorders; veteran
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic | interventions — Dexamethasone; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Dexamethasone (Experimental): Dexamethasone (oral)
  Interventions: Drug: Dexamethasone
- Arm 2: Placebo (Placebo Comparator): Placebo (inactive)
  Interventions: Drug: Placebo (sugar pill)

INTERVENTIONS:
Drug: Dexamethasone — anti-inflammatory adrenocortical steroid The following dose schedule will be given: 0.15mg/kg (based on body weight) every 7 days for 4 consecutive weeks
  Arms: Arm 1: Dexamethasone
Drug: Placebo (sugar pill) — inactive
  Arms: Arm 2: Placebo

SUMMARY:
The purpose of this study is to examine the effects of glucocorticoid administration following traumatic memory reactivation on psychiatric symptoms in veterans with combat-related PTSD, in addition to examining the effects of glucocorticoid administration following traumatic memory reactivation on physiological responses to veteran's personal combat memories. The following hypotheses will be tested:

1. Subjects who receive an exogenous glucocorticoid after traumatic memory reactivation will demonstrate fewer PTSD and depression symptoms one week later, compared to those who receive a placebo after traumatic memory reactivation.
2. The glucocorticoid reduction effects will be cumulative; that is, reduction will persist, and further post-reactivation glucocorticoid administration will further reduce symptoms
3. Decreases in PTSD and depression symptoms will persist at 1, 3, and 6 months for subjects receiving an exogenous glucocorticoid compared to those subjects receiving placebo
4. Subjects who receive an exogenous glucocorticoid after traumatic memory reactivation will demonstrate decreased physiological responses one week later, compared to those who receive a placebo after traumatic memory reactivation.
5. As with the psychological measures, suppression of the physiological measures will demonstrate both persistence over time and accumulation with subsequent post-reactivation glucocorticoid administration.

DETAILED DESCRIPTION:
Background information and related research:

Post-traumatic stress disorder (PTSD) is characterized, among other things, by intrusive memories in the form of unwanted images, nightmares, and flashbacks. These memories are associated with intense distress and involve excessive physiological and psychological responses to fear associated stimuli. Prevalence rates of combat-related PTSD are increasing due to Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) deployments, with the estimated risk for PTSD from service in the Iraq War at 18%, and 11% for Afghanistan.

According to the Pentagon's own mental health taskforce, 38% of soldiers, 31% of marines, 49% of National Guard members, and 43% of marine reservists have shown symptoms of post-traumatic stress disorder or other psychological problems within three months of returning from active duty. Estimates from the National Center on PTSD suggest that 40% of OEF/OIF troops may have or will acquire PTSD. The Department of Defense (DoD) reports that 22% of OEF/OIF troops have been flagged for PTSD and referred for follow-up care, and records indicate that over 39,000 OEF/OIF vets had been treated for PTSD as of December, 2006.

Current research efforts are exploring the underlying neurochemical changes associated with PTSD. Recently, these efforts have focused on the prevention of PTSD in persons exposed to trauma by administration of medication to affect the underlying neurochemical processes. For example, preliminary evidence suggests that interference with consolidation of trauma-related memories using the beta-antagonist, propranalol, may prevent PTSD in humans with recent traumas. However, given that as much as 90% of the US population is exposed to at least one traumatic event during their lifetime, the utility of this treatment is limited by the logistical problems of treating everyone at risk for developing PTSD after a trauma. To date, there are very few systematic studies on humans that focus on changing the underlying traumatic memory once PTSD has been established.

The trauma experience is initially stored in short-term memory, then consolidated into long-term memory. However, the long-term stability conferred by the consolidation process undergoes a period of labiality as follows. Each time a consolidated memory is activated, the memory trace becomes newly labile and must be consolidated again to remain in long-term memory. This process is called reconsolidation. Reconsolidation therefore offers a biologic window during which long-term memories can be disrupted. Preclinical studies have begun to unravel the biological changes that underlie these processes. Both pharmacological agents, including glucocorticoids, and protein synthesis inhibitors can interfere with memory consolidation and reconsolidation. Endogenously produced stress-hormones, or glucocorticoids, enhance consolidation for emotionally-arousing experiences, but these effects are dependent on dose, aversiveness of task, and timing of hormone administration. Conversely, glucocorticoids appear to impair the retrieval of memories of aversive experiences.10 Recent data also suggest that glucocorticoids enhance extinction of traumatic memories.

Preclinical work in our laboratory at the UT Southwestern Medical Center has established that corticosterone can dose-dependently reduce an established fear memory in rodents. In this study, mice were trained to associate foot-shock with a specific training context to induce fear memory. When this fear memory was reactivated by the contextual stimulus and then followed by glucocorticoid administration, subsequent reactivation of the fear memory produced significantly less fear responses relative to mice administered saline after memory reactivation. After only one pairing of reactivation and glucocorticoid, this effect was reversible with a subthreshold reminder shock and was transient, indicating that the effect of glucocorticoids was on the extinction process. These results strongly suggested glucocorticoid treatment paired with therapeutic traumatic memory reactivation as a specific therapy for PTSD in humans and directly informed our pilot studies in PTSD patients.

ELIGIBILITY:
Inclusion Criteria:

* male veterans enrolled to receive care through the VA North Texas Healthcare System
* diagnosis of combat-related PTSD

Exclusion Criteria:

* Hypersensitivity to dexamethasone
* Current use of steroids
* Current psychosis
* Organic Brain Damage
* Current major depressive disorder with melancholic features
* Substance dependence in the last 3 months
* Prominent suicidal or homicidal features
* Medical conditions: diabetes, uncontrolled hypertension, severe congestive heart failure, hepatic failure, or any other contraindicated medical condition (such as HPA Axis disease, Addison's Disease or Cushing's Disease).
* Veterans taking medication with established drug interactions with dexamethasone

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2010-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alina M Suris, PhD, Principal Investigator — VA North Texas Health Care System, Dallas
Locations (1):
- VA North Texas Health Care System, Dallas, Dallas, Texas, United States

REFERENCES:
- [Derived] Suris A, Holliday R, Adinoff B, Holder N, North CS. Facilitating Fear-Based Memory Extinction With Dexamethasone: A Randomized Controlled Trial in Male Veterans With Combat-Related PTSD. Psychiatry. 2017 Winter;80(4):399-410. doi: 10.1080/00332747.2017.1286892. PMID 29466111

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 67 participants excluded from initial recruitment sample for the following reasons: baseline assessment inclusion criteria not met (n = 18), declined enrollment post-consent (n = 1), exclusion criteria met (n = 26), lost to follow-up (n = 24).
Period: Overall Study
Arm/Group | Arm 1: Dexamethasone | Arm 2: Placebo
Started | 33 | 29
Completed | 22 | 21
Not Completed | 11 | 8

BASELINE CHARACTERISTICS:
Population: Male veterans with combat-related PTSD
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Dexamethasone | Arm 2: Placebo | Total
Number analyzed (Participants) | 33 | 29 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.91 (11.74) | 41.34 (13.97) | 37.92 (12.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 33 | 29 | 62
Race/Ethnicity, Customized [Number; unit: participants]
  White, non-Hispanic | 19 | 17 | 36
  Black, non-Hispanic | 11 | 7 | 18
  White, Hispanic | 1 | 1 | 2
  Other | 1 | 4 | 5
  Declined to state | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 33 | 29 | 62

OUTCOME MEASURES:

1. Primary Outcome: PTSD Checklist (PCL). A Self-report, Face Valid Measure of PTSD Symptoms Over a 1 Week Time Period
Description: The PCL is a 17-item measure of PTSD symptom severity with a range from 17-85. Each item is rated from 1-5 with higher scores are indicative of higher symptom severity. Scores of the 17 items are summed in order to generate the total score.
Time Frame: This measure will be administered at all study visits: Baseline, 1 month, 3 months, and 6 months follow up.
Population: Male veterans with combat-related PTSD
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Dexamethasone | Arm 2: Placebo
Number analyzed (Participants) | 33 | 29
units on a scale
  Baseline | 55.76 (10.17) | 54.83 (12.19)
  1-month follow up | 50.14 (13.35) | 51.57 (11.36)
  3-month follow up | 45.45 (13.80) | 51.89 (12.39)
  6-month follow up | 58.57 (13.72) | 48.17 (12.53)

2. Secondary Outcome: Quick Inventory of Depressive Symptomatology- Self Report (QIDS-SR). Because Depression Can be Comorbid With PTSD (70% Comorbidity Found in Pilot Sample), This Assessment Will be Used to Measure Depressive Symptoms Over a 1 Week Timeframe
Description: The QIDS-SR is a 16-item measure of depression symptom severity with a range from 0-27. Each item is rated from 0-3 with higher scores are indicative of higher symptom severity. Scores of the items are aggregated (with the highest score on overlapping items chosen; e.g., sleep disturbances, changes in eating) to generate the total score..
Time Frame: This measure will be administered at all study visits: Baseline, 1 month, 3 months, and 6 months follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Dexamethasone | Arm 2: Placebo
Number analyzed (Participants) | 33 | 29
units on a scale
  Baseline | 13.55 (4.59) | 12.86 (3.36)
  1-month follow up | 10.68 (4.36) | 10.71 (3.54)
  3-month follow up | 11.38 (5.12) | 11.32 (3.59)
  6-month follow up | 11.00 (5.62) | 10.33 (3.68)

ADVERSE EVENTS:
Arm/Group | Arm 1: Dexamethasone | Arm 2: Placebo
Serious Adverse Events (participants affected / at risk) | 1/33 | 0/29
Other Adverse Events (participants affected / at risk) | 0/33 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Dexamethasone (N=33) | Arm 2: Placebo (N=29)
Presented to ER with swelling in leg (Infections and infestations) | 1 (1) | 0 (0) — Diagnosed with cellulitis at the ER. Determined to be possibly related due to potential immunosuppression from study medication. Reported to IRB and informed consent was updated accordingly.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No